CLINICAL TRIAL: NCT05755191
Title: A Phase 1, Single and Multiple Ascending Dose and Food Effect Study of NEU-411 Administered Orally to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics in Healthy Subjects
Brief Title: A Study to Assess NEU-411 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neuron23 Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NEU-411-PD101
Record Dates: First submitted 2023-02-22; First posted 2023-03-06 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- NEU-411 (Experimental): Part A: Single-ascending dose cohorts; food effect; Part B: Multiple-ascending dose cohorts (7 days)
  Interventions: Drug: NEU-411
- Placebo (Placebo Comparator): Part A: Single-ascending dose cohorts; food effect; Part B: Multiple-ascending dose cohorts (7 days)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NEU-411 — Oral Doses
  Arms: NEU-411
Drug: Placebo — Oral Doses
  Arms: Placebo

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, single ascending dose (SAD), food effect (FE),multiple ascending dose (MAD), drug-drug interaction study, and bioavailability - bio-equivalence study of orally administered NEU-411 in healthy subjects

DETAILED DESCRIPTION:
Up to five (5) single-ascending oral doses will be administered to 40 healthy adult male or female subjects (aged 18-80 years, inclusive). Escalation to the next higher dose level may occur only after evaluation of the safety and PK results of the previous dose level (at least 6 evaluable subjects). Within each cohort, 6 subjects will receive one dose of NEU-411, and 2 subjects will receive one dose of matching placebo. Dose levels may be revised based on available safety and PK data.

Food effect will evaluate approximately 8 subjects in a fasted versus fed state.

Multiple ascending oral doses will be administered up to 24 healthy subjects (aged 18 - 80 years, inclusive) in 3 sequential dosing groups (8 subjects in each dosing group). Six (6) subjects will receive NEU-411 and two (2) subjects will receive matching placebo in each dosing group (cohort) for 7 days. Escalation to the next higher dose level may occur only after evaluation of the safety and PK results of the previous dose level (at least 6 evaluable subjects). Dose levels may be revised based on available safety and PD data.

Multiple oral dosing will be administered in up to 39 healthy subjects in 3 sequential dosing groups (13 subjects across 3 dosing groups) over 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects for standard cohorts must be 18-80 years, inclusive, at the time of signing the informed consent;
* Subjects who are in good general health with no clinically relevant abnormalities based on the medical history, physical examinations, neurological examinations, clinical laboratory evaluations (hematology and clinical chemistry)
* Subjects who have a body mass index (BMI) of 18-32 kg/m2(inclusive);
* Male subjects are eligible to participate if they are rendered surgically sterile (at least 6 months), or agree to the following during the study and for at least 30 days after the last dose of study drug:
* Refrain from donating sperm;

AND, either:

Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent; OR Agree to use a male condom (contraception/barrier) and should also be advised of the benefit for a female partner to use an acceptable, highly effective method of contraception as a condom may break or leak when having sexual intercourse;

• Female subjects are eligible to participate if they are not pregnant or breastfeeding, subject to one of the following:

* Women of childbearing potential (WOCBP), defined as women physiologically capable of becoming pregnant, must have a negative serum pregnancy test at the Screening visit and a negative urine pregnancy test on Day -1; WOCBP must agree to use an acceptable, highly effective contraceptive method from Screening until 30 days after the last dose of study treatment (see Section 11.3); OR
* Menopausal women must have an elevated serum follicle-stimulating hormone level (FSH) level at Screening; if the FSH is not elevated, they are considered to be of childbearing potential (unless permanently sterile) and must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day -1

Exclusion Criteria:

* History of clinically significant hematological, renal, pancreatic, gastrointestinal, hepatic, cardiovascular, metabolic, endocrine, immunological, allergic disease, or other major disorders
* History of clinically significant abnormal chest x-ray
* Clinically significant neurologic disorder
* Contraindications to undergo a lumbar puncture (only for subjects participating in the MAD)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2023-05-13 (Actual); Primary Completion 2024-06-03 (Actual); Study Completion 2024-06-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of single dosing, food effect and multiple oral doses of NEU-411 in healthy subjects | Up to 7 days of dosing
  Incidence of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
PK parameter | Up to 7 days of dosing
  The maximum concentration (Cmax) at steady state in plasma
PK parameter | Up to 7 days of dosing
  The area under the concentration-time curve from zero to infinity (AUC0-inf) in plasma
PK parameter | Up to 7 days of dosing
  The time to reach maximum concentration (tmax) in plasma
PK parameter | Up to 7 days of dosing
  Area under the concentration-time curve from time zero to the time of last quantifiable concentration (AUC[0-last]) in plasma
PK parameter | Up to 7 days of dosing
  Apparent terminal elimination half-life (t1/2) in plasma
PK parameter | Up to 7 days of dosing
  The terminal elimination rate constant (λZ) with the respective half-life (t½) in plasma
PK parameter | Up to 7 days of dosing
  The oral clearance (CL/F)
PK parameter | Up to 7 days of dosing
  The volume of distribution (Vd/F)
PK parameter | Up to 7 days of dosing
  The area under the concentration-time curve over a dosing interval (AUC0-τ) in plasma (multiple dosing only)

CONTACTS AND LOCATIONS:
Locations (1):
- New Zealand Clinical Research, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No